CLINICAL TRIAL: NCT05572125
Title: Oral Iron Therapy in Erythropoietic Protoporphyria
Brief Title: Iron Therapy in Erythropoietic Protoporphyria
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Alfred Benzon Foundation (Unknown)
Responsible Party: Principal Investigator, Ida M. Heerfordt, Principal Investigator, Bispebjerg Hospital
Other Study IDs: Iron
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Erythropoietic Protoporphyria; Iron-deficiency
MeSH Terms: conditions — Protoporphyria, Erythropoietic; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Giving oral iron to patients with erythropoietic protoporphyria (EPP) who is iron deficient is thought to be beneficial. This is, however, not well documented. The purpose of this study is to investigate the effect and safety of oral iron in patients with EPP who is taking iron tablets due to iron deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with EPP
* Taking standard dose of iron tablets due to iron deficiency

Exclusion Criteria:

* Pregnant
* Lactating

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with EPP taking oral iron tablets due to iron deficiency
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Change in erythrocyte protoporphyrin concentration | Before treatment and after 6-8 weeks of treatment

SECONDARY OUTCOMES:
Change in hemoglobin and iron parameters | Before treatment and after 6-8 weeks of treatment
Adverse event | 6-8 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark